CLINICAL TRIAL: NCT06762002
Title: Impaired Type I IFN Immunity Due to Autoantibodies or a Genetic Defect: a Prospective National Cohort
Acronym: COVIFERON
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C22-73; 2023-A02663-42 (Other: ANSM ID-RCB)
Record Dates: First submitted 2024-11-14; First posted 2025-01-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-12

CONDITIONS: Immunology; Allergy; Genetic Diseases; Infectious Diseases
Keywords: covid-19; auto-immunity; Type I interferon; kinetics; infectious diseases
MeSH Terms: conditions — Hypersensitivity; Genetic Diseases, Inborn; Communicable Diseases; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood samples for:
  * full blood cell count;
  * classical autoimmune investigations (anti-nuclear, anti-ENA, native anti-DNA, anti- thyroid antibodies, rheumatoid factor);
  * immunophenotyping;
  * auto-Abs against type I IFNs, other cytokines, or other target proteins (dosage and neutralization activity);
  * Genetic explorations by whole-exome or whole-genome sequencing;
  * Biobanking (DNA, plasma/sera; cryopreserved peripheral blood mononuclear cells (PBMCs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with auto-Abs against type I IFNs or inborn errors of immunity: The study examines how autoantibodies (auto-Abs) against type I interferons (IFNs) and inborn errors of immunity affect susceptibility to infectious diseases, especially COVID-19. Individuals with auto-Abs against type I IFNs have impaired immune responses to viral infections, putting them at higher risk for severe COVID-19, leading to worse outcomes like pneumonia or cytokine storms. Those with inborn errors of immunity have genetic defects that weaken immune function, increasing vulnerability to infections, including COVID-19. The study compares these groups to understand immune dysfunctions and identify potential therapeutic targets.
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — After signature of consent form,blood samples will be collected for full blood cell count;classical autoimmune investigations, immunophenotyping;auto-Abs against type IIFNs, other cytokines, or other target proteins ,Genetic explorations by whole-exome or whole-genome sequencing;Biobanking

SUMMARY:
The major role of human genetic factors in the immune response to infections is now well established, particularly for viral infections. In the context of the COVID-19 pandemic, the following results have identified 1) several inborn errors of immunity (IEI) affecting the response or production of type I interferons (type I IFNs) in around 4% of adult patients with severe clinical disease, and 2) the presence of type I IFN-neutralizing autoantibodies (auto-Abs) in around 15% of severe cases, and 20% of deaths. The investigators would like to carry out a longitudinal immunological and clinical follow-up study on a prospective cohort of patients with either a genetic defect affecting the type I IFN-dependent immune response, or anti-IFN-I auto-Abs, to monitor the incidence of infectious and/or autoimmune events in these individuals, the evolution of neutralizing power, and the kinetics of auto-Abs. This should lead to a better understanding of the prevention and management of these patients.

The research design is a national multicenter prospective cohort of adults with 1) anti-IFN-I auto-Abs or 2) IEI- IFN-I, with follow-up from 1 to 4 years. These individuals may be: 1) patients who have or have had clinical disease (related to COVID-19, other viral infections, autoimmune disorders); or 2) "healthy" participants (e.g. blood donors, relatives of an IEI patient).

Follow-up will include:

* yearly visits to the Clinical Investigation Center (CIC) or a clinical department with blood sampling;
* specific visit in case of hospitalization for infectious events or adverse effects of vaccination, exacerbation or new diagnosis of auto-immune disease, new diagnosis of cancer, or SARS-CoV-2 infection whether or not patients are admitted to hospital, with blood sampling.

In addition, a retrospective "passive" follow-up will be implemented through matching with the data from the SNDS (National Health Data System), in order to collect clinical events of and healthcare resource consumption. Moreover, matching with controls adults from the national CONSTANCES cohort, not carrying auto-Abs against type I IFNs nor IEI-IFN-I, will be performed. (ratio 3:1; matching on age (+/- 5 years), gender and geographic region of recruitment). Individuals under long-lasting immunosuppressive or immunomodulatory drugs will not be eligible. Follow-up of controls, which will be carried out as part of the CONSTANCES cohort, will include web-based questionnaires, every 12 months, in addition to linking with SNDS data as already done in this cohort.

Inclusion visit:

After signing the consent form, the following tests will be performed:

* Demographic characteristics (sex, age, country of birth)
* Medical history from participant and family member(s) including infectious and auto-immune diseases, cancers and vaccination status and side effects
* Blood samples for:

  * full blood cell count;
  * classical autoimmune investigations (anti-nuclear, anti-ENA, native anti-DNA, anti- thyroid antibodies, rheumatoid factor);
  * immunophenotyping*;
  * auto-Abs against type I IFNs, other cytokines*, or other target proteins* (dosage and neutralization activity);
  * Genetic explorations by whole-exome or whole-genome sequencing*;
  * Biobanking (DNA, plasma/sera; cryopreserved peripheral blood mononuclear cells (PBMCs).

    * these biological analyses will be carried out as part of dedicated COVIFERON RHU5 workpackages.

In addition, vaccination against SARS-CoV-2 and influenza will be offered to these subjects as a priority, as part of their usual care.

Follow-up visits :

Annual visits to the CIC :

* Medical history since last visit, including infectious, auto-immune and oncologic events, vaccination status and side effects
* Blood samples for:

  * full blood cell count;
  * classical autoimmune investigation (anti-nuclear, anti-ENA, native anti- DNA, anti-thyroid antibodies, rheumatoid factor);
  * immunophenotyping;
  * Auto-Abs against type I IFNs, other cytokines, or other target proteins (dosage and neutralization)
  * Biobanking (DNA, plasma, cryopreserved peripheral blood mononuclear cells (PBMCs))

Additional specific visit in the event of a clinical event of interest, at any time during follow-up:

* In case of SARS-CoV-2 infection, whatever the severity of the disease: blood sampling for determination and neutralization of type I anti-IFN autoAbs, CBC, and biobanking (plasma and PBMC) and teleconsultation with the CIC in charge of patients, as soon as possible.
* In the event of hospitalization for infectious events or exacerbation or new diagnosis of an auto-immune disease: blood sampling for determination and neutralization of anti-IFN-I autoAbs, CBC, and biobanking (plasma and PBMCs) and collection of the hospitalization report in the case report form on a dedicated page.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* History of carrying 1) auto-Abs against type I IFNs or 2) IEI impairing the response to, or the production of, type I IFNs (IFN-I-IEI)
* Affiliated to social security
* Written informed consent

Exclusion Criteria:

* Participation to an interventional clinical trial on a pharmacological treatment
* Clinical condition leading to life expectancy less than 1 year
* Subject to a legal protection measure (safeguard of justice, curatorship, tutorship)
* Individuals deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with auto-Abs against IFN-I or an IEI-IFN-I who: 1) either have or have had a clinical disease (COVID-19 related, other viral infections, adverse effect of vaccination, auto-immune disorders); or 2) are healthy (e.g. blood donor, relatives of a participant).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
primary endpoint n°1 : quantitative dosage of auto-Abs against type I IFNs | year 0, year 1, year 2 and year 3
  Method: Quantitative trait will be measured by Gyros using commercially available internal control antibodies.
primary endpoint n°2 : neutralization capacity evaluation of auto-Abs against type I IFNs | year 0, year 1, year 2 and year 3
  The neutralization capacity will be performed as previously reported using an in vitro luciferase system in HEK293 cells

SECONDARY OUTCOMES:
Cumulative incidence of clinical events of interest, i.e. infectious events, autoimmune diseases or cancers | Year 0, year 1, year 2 and year 3
  Method: annual medical visits, SNDS (PMSI, DCIR). Incidence density rate is defined as the number of newly disease individuals on the sum of time periods for all disease-free individual-at-risk
Clinical and biological factors associated with clinical outcomes | Year 0, year 1, year 2 and year 3
  the potential predictor variables will be assessed by bivariate logistic regressions where occurrence of clinical events is the variable to be explained. Factors associated with a p-value less than 0.20 will be included in the multivariate logistic model. Backward selection on pvalue will be applied. Internal validity of the final model will be estimated by cross-validation (Leave-One-Out Cross-Validation method). Discrimination will be assessed by the area under the ROC curve and its 95% confidence interval.
Cumulative incidence of the same clinical events of interest, in control participants who are negative for auto-Abs, matched by age and sex followed through the large CONSTANCES cohort | Year 0, year 1, year 2 and year 3
  Cumulative incidence of the same clinical events of interest, in control participants who are negative for auto-Abs, matched by age and sex followed through the large CONSTANCES cohort (Constances database), and its 95% confidence interval: Incidence density rate is defined as the number of newly disease individuals on the sum of time periods for all disease-free individual-at-risk.
Genetic factors associated with the development of auto-Abs against type I IFNs | Year 0, year 1, year 2 and year 3
  searching for homozygous deletions using in-house HMZDelFinder-opt method of imagine institue
Genetic factors associated with the development of auto-Abs against type I IFNs | year 0, year 1, year 2 and year 3
  Searching for rare candidate coding variants in patients by following an optimal filtering strategy that imagine have optimized over the last 10 years based on multiple variant-level and gene-level criteria to select the candidate variants
Genetic factors associated with the development of auto-Abs against type I IFNs | year 0, year 1, year 2 and year 3
  Using gene-level criteria to select candidate variants such as the negative selection level measured by the CoNeS approach.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Cic Lille, Lille
  - LYON HCL, Lyon
  - Cic Montpellier, Montpellier
  - Cic Bichat, Paris
  - Cic Creteil, Paris
  - Cic La Salpetriere, Paris
  - Cic Necker, Paris
  - Cic St Louis, Paris
  - Cic Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bastard P, Gervais A, Le Voyer T, Rosain J, Philippot Q, Manry J, Michailidis E, Hoffmann HH, Eto S, Garcia-Prat M, Bizien L, Parra-Martinez A, Yang R, Haljasmagi L, Migaud M, Sarekannu K, Maslovskaja J, de Prost N, Tandjaoui-Lambiotte Y, Luyt CE, Amador-Borrero B, Gaudet A, Poissy J, Morel P, Richard P, Cognasse F, Troya J, Trouillet-Assant S, Belot A, Saker K, Garcon P, Riviere JG, Lagier JC, Gentile S, Rosen LB, Shaw E, Morio T, Tanaka J, Dalmau D, Tharaux PL, Sene D, Stepanian A, Megarbane B, Triantafyllia V, Fekkar A, Heath JR, Franco JL, Anaya JM, Sole-Violan J, Imberti L, Biondi A, Bonfanti P, Castagnoli R, Delmonte OM, Zhang Y, Snow AL, Holland SM, Biggs C, Moncada-Velez M, Arias AA, Lorenzo L, Boucherit S, Coulibaly B, Anglicheau D, Planas AM, Haerynck F, Duvlis S, Nussbaum RL, Ozcelik T, Keles S, Bousfiha AA, El Bakkouri J, Ramirez-Santana C, Paul S, Pan-Hammarstrom Q, Hammarstrom L, Dupont A, Kurolap A, Metz CN, Aiuti A, Casari G, Lampasona V, Ciceri F, Barreiros LA, Dominguez-Garrido E, Vidigal M, Zatz M, van de Beek D, Sahanic S, Tancevski I, Stepanovskyy Y, Boyarchuk O, Nukui Y, Tsumura M, Vidaur L, Tangye SG, Burrel S, Duffy D, Quintana-Murci L, Klocperk A, Kann NY, Shcherbina A, Lau YL, Leung D, Coulongeat M, Marlet J, Koning R, Reyes LF, Chauvineau-Grenier A, Venet F, Monneret G, Nussenzweig MC, Arrestier R, Boudhabhay I, Baris-Feldman H, Hagin D, Wauters J, Meyts I, Dyer AH, Kennelly SP, Bourke NM, Halwani R, Sharif-Askari NS, Dorgham K, Sallette J, Sedkaoui SM, AlKhater S, Rigo-Bonnin R, Morandeira F, Roussel L, Vinh DC, Ostrowski SR, Condino-Neto A, Prando C, Bonradenko A, Spaan AN, Gilardin L, Fellay J, Lyonnet S, Bilguvar K, Lifton RP, Mane S; HGID Lab; COVID Clinicians; COVID-STORM Clinicians; NIAID Immune Response to COVID Group; NH-COVAIR Study Group; Danish CHGE; Danish Blood Donor Study; St. James's Hospital; SARS CoV2 Interest group; French COVID Cohort Study Group; Imagine COVID-Group; Milieu Interieur Consortium; CoV-Contact Cohort; Amsterdam UMC Covid-19; Biobank Investigators; COVID Human Genetic Effort; CONSTANCES cohort; 3C-Dijon Study; Cerba Health-Care; Etablissement du Sang study group; Anderson MS, Boisson B, Beziat V, Zhang SY, Vandreakos E, Hermine O, Pujol A, Peterson P, Mogensen TH, Rowen L, Mond J, Debette S, de Lamballerie X, Duval X, Mentre F, Zins M, Soler-Palacin P, Colobran R, Gorochov G, Solanich X, Susen S, Martinez-Picado J, Raoult D, Vasse M, Gregersen PK, Piemonti L, Rodriguez-Gallego C, Notarangelo LD, Su HC, Kisand K, Okada S, Puel A, Jouanguy E, Rice CM, Tiberghien P, Zhang Q, Cobat A, Abel L, Casanova JL. Autoantibodies neutralizing type I IFNs are present in ~4% of uninfected individuals over 70 years old and account for ~20% of COVID-19 deaths. Sci Immunol. 2021 Aug 19;6(62):eabl4340. doi: 10.1126/sciimmunol.abl4340. PMID 34413139
- [Background] Zhang Q, Bastard P, Liu Z, Le Pen J, Moncada-Velez M, Chen J, Ogishi M, Sabli IKD, Hodeib S, Korol C, Rosain J, Bilguvar K, Ye J, Bolze A, Bigio B, Yang R, Arias AA, Zhou Q, Zhang Y, Onodi F, Korniotis S, Karpf L, Philippot Q, Chbihi M, Bonnet-Madin L, Dorgham K, Smith N, Schneider WM, Razooky BS, Hoffmann HH, Michailidis E, Moens L, Han JE, Lorenzo L, Bizien L, Meade P, Neehus AL, Ugurbil AC, Corneau A, Kerner G, Zhang P, Rapaport F, Seeleuthner Y, Manry J, Masson C, Schmitt Y, Schluter A, Le Voyer T, Khan T, Li J, Fellay J, Roussel L, Shahrooei M, Alosaimi MF, Mansouri D, Al-Saud H, Al-Mulla F, Almourfi F, Al-Muhsen SZ, Alsohime F, Al Turki S, Hasanato R, van de Beek D, Biondi A, Bettini LR, D'Angio' M, Bonfanti P, Imberti L, Sottini A, Paghera S, Quiros-Roldan E, Rossi C, Oler AJ, Tompkins MF, Alba C, Vandernoot I, Goffard JC, Smits G, Migeotte I, Haerynck F, Soler-Palacin P, Martin-Nalda A, Colobran R, Morange PE, Keles S, Colkesen F, Ozcelik T, Yasar KK, Senoglu S, Karabela SN, Rodriguez-Gallego C, Novelli G, Hraiech S, Tandjaoui-Lambiotte Y, Duval X, Laouenan C; COVID-STORM Clinicians; COVID Clinicians; Imagine COVID Group; French COVID Cohort Study Group; CoV-Contact Cohort; Amsterdam UMC Covid-19 Biobank; COVID Human Genetic Effort; NIAID-USUHS/TAGC COVID Immunity Group; Snow AL, Dalgard CL, Milner JD, Vinh DC, Mogensen TH, Marr N, Spaan AN, Boisson B, Boisson-Dupuis S, Bustamante J, Puel A, Ciancanelli MJ, Meyts I, Maniatis T, Soumelis V, Amara A, Nussenzweig M, Garcia-Sastre A, Krammer F, Pujol A, Duffy D, Lifton RP, Zhang SY, Gorochov G, Beziat V, Jouanguy E, Sancho-Shimizu V, Rice CM, Abel L, Notarangelo LD, Cobat A, Su HC, Casanova JL. Inborn errors of type I IFN immunity in patients with life-threatening COVID-19. Science. 2020 Oct 23;370(6515):eabd4570. doi: 10.1126/science.abd4570. Epub 2020 Sep 24. PMID 32972995
- [Background] Bastard P, Rosen LB, Zhang Q, Michailidis E, Hoffmann HH, Zhang Y, Dorgham K, Philippot Q, Rosain J, Beziat V, Manry J, Shaw E, Haljasmagi L, Peterson P, Lorenzo L, Bizien L, Trouillet-Assant S, Dobbs K, de Jesus AA, Belot A, Kallaste A, Catherinot E, Tandjaoui-Lambiotte Y, Le Pen J, Kerner G, Bigio B, Seeleuthner Y, Yang R, Bolze A, Spaan AN, Delmonte OM, Abers MS, Aiuti A, Casari G, Lampasona V, Piemonti L, Ciceri F, Bilguvar K, Lifton RP, Vasse M, Smadja DM, Migaud M, Hadjadj J, Terrier B, Duffy D, Quintana-Murci L, van de Beek D, Roussel L, Vinh DC, Tangye SG, Haerynck F, Dalmau D, Martinez-Picado J, Brodin P, Nussenzweig MC, Boisson-Dupuis S, Rodriguez-Gallego C, Vogt G, Mogensen TH, Oler AJ, Gu J, Burbelo PD, Cohen JI, Biondi A, Bettini LR, D'Angio M, Bonfanti P, Rossignol P, Mayaux J, Rieux-Laucat F, Husebye ES, Fusco F, Ursini MV, Imberti L, Sottini A, Paghera S, Quiros-Roldan E, Rossi C, Castagnoli R, Montagna D, Licari A, Marseglia GL, Duval X, Ghosn J; HGID Lab; NIAID-USUHS Immune Response to COVID Group; COVID Clinicians; COVID-STORM Clinicians; Imagine COVID Group; French COVID Cohort Study Group; Milieu Interieur Consortium; CoV-Contact Cohort; Amsterdam UMC Covid-19 Biobank; COVID Human Genetic Effort; Tsang JS, Goldbach-Mansky R, Kisand K, Lionakis MS, Puel A, Zhang SY, Holland SM, Gorochov G, Jouanguy E, Rice CM, Cobat A, Notarangelo LD, Abel L, Su HC, Casanova JL. Autoantibodies against type I IFNs in patients with life-threatening COVID-19. Science. 2020 Oct 23;370(6515):eabd4585. doi: 10.1126/science.abd4585. Epub 2020 Sep 24. PMID 32972996